CLINICAL TRIAL: NCT01544920
Title: A Phase 3, Safety and Efficacy Study of Boceprevir/Peginterferon Alfa-2a/Ribavirin in Chronic HCV Genotype 1 IL28B CC Subjects
Brief Title: Safety and Efficacy of Boceprevir/Peginterferon Alfa-2a/Ribavirin in Interleukin-28B CC Allele-Positive Chronic Hepatitis C Virus (HCV) Genotype 1 Participants (P07755)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07755; 2011-001345-32 (EudraCT Number); MK-3034-040 (Other: Merck); CTRI/2012/12/003200 (Registry Identifier: CTRI); PHRR131022-000133 (Registry Identifier: PHRR)
Record Dates: First submitted 2012-02-28; First posted 2012-03-06 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: peg-IFN + RBV (Active Comparator): Participants received an initial 4 week lead-in of peg-IFN + RBV. Following HCV RNA analysis at Week 4, participants with undetectable HCV RNA received open label peg-IFN + RBV for an additional 18 weeks (total of 24 weeks of peg-IFN/RBV therapy) [Arm 1a]. Participants with detectable HCV RNA at Week 4 had BOC added to the peg-IFN + RBV regimen at Week 6 and then followed the Response Guided Therapy (RGT) regimen for BOC + peg-IFN + RBV [Arm 1b].
  Interventions: Biological: peg-Interferon alfa-2a; Drug: Ribavirin; Drug: Boceprevir
- Arm 2: BOC + peg-IFN + RBV (Experimental): Participants received an initial 4-week lead-in of peg-IFN + RBV. Following HCV RNA analysis at Week 4, all participants had BOC added to the peg-IFN + RBV regimen at Week 6 regardless of HCV RNA levels. Participants who had undetectable HCV RNA at Week 4 continued on the BOC + peg-IFN + RBV regimen for an additional 20 weeks (total of 24 weeks of BOC + peg-IFN + RBV therapy) [Arm 2a]. Participants with detectable HCV RNA at Week 4 followed the RGT regimen for BOC + peg-IFN + RBV [Arm 2b].
  Interventions: Biological: peg-Interferon alfa-2a; Drug: Ribavirin; Drug: Boceprevir

INTERVENTIONS:
Biological: peg-Interferon alfa-2a — peg-IFN (180 ug) was taken once weekly via subcutaneous injection.
  Other Names: Pegasys™; SCH 054031
Drug: Ribavirin — RBV 200 mg tablets taken by mouth at a total daily dose of 1,000 mg (body weight <75 kilograms [kg]) or 1,200 mg (body weight ≥75 kg) with total daily dose divided into 2 dosings.
  Other Names: Rebetol™; 018908
Drug: Boceprevir — Four 200 mg BOC capsules taken three times a day by mouth for a total daily dose of 2,400 mg.
  Other Names: SCH 503034; Victrelis™

SUMMARY:
The primary purpose of this study is to compare the efficacy of two boceprevir (BOC)-containing therapeutic regimens in the treatment of naïve participants with chronic hepatitis C virus (HCV) genotype 1 who have the IL28B CC allele.

The regimens differ in the treatment for participants who achieve undetectable HCV ribonucleic acid (RNA) at the end of the peginterferon alfa-2a (peg-IFN) plus ribavirin (RBV) 4 week lead-in. Participants receive either peg-IFN + RBV (Arm 1) or BOC + peg-IFN + RBV (Arm 2). The hypothesis is that Arm 2 is noninferior to Arm 1 in the proportion of participants with undetectable HCV RNA at Follow-Up (FU) Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥ 40 kg and ≤ 125 kg.
* Documented CHC genotype 1 with HCV RNA ≥10,000 International Units (IU)/mL
* Has IL-28B CC allele gene
* Has had a liver biopsy without evidence of cirrhosis and hepatocellular carcinoma (non-invasive fibroscan and Fibrotest can also be used for staging of liver disease).

Exclusion Criteria:

* Co-infection with the human immunodeficiency virus (HIV) or hepatitis B virus (Hepatitis B surface antigen [HBsAg] or HIV positive).
* Previously treated with an interferon and ribavirin regimen or HCV direct acting antiviral regimen.
* Treatment for hepatitis C with any investigational medication, or prior treatments with herbal remedies with known hepatotoxicity
* Receiving any medication(s) within 2 weeks prior to the Day 1 visit that are highly dependent on Cytochrome P450 3A4 (CYP3A4/5) for clearance, and for which elevated plasma concentrations could be associated with serious and/or life-threatening events
* Participation in any other clinical trial within 30 days of the screening visit in this trial or intention to participate in another clinical trial during participation in this trial.
* Evidence of decompensated liver disease or hepatocellular carcinoma (HCC)
* Is diabetic and/or hypertensive with significant retinopathy
* Has any known medical condition that could interfere with the participation in and completion of the trial including immunologically-mediated disease, chronic pulmonary disease, or current or history of any clinically significant cardiac abnormalities/dysfunction.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years
* Hemoglobin <12 g/dL for females and <13 g/dL for males
* Neutrophils <1,500/mm^3, or <1,200/mm^3 for participants of African descent
* Platelets <150,000/mm^3
* Direct bilirubin >1.5 x upper limit of normal (ULN) of the laboratory reference range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2015-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Peg-IFN + RBV | Arm 2: BOC + Peg-IFN + RBV
Started | 368 | 369
Completed | 349 | 346
Not Completed | 19 | 23
Not completed — Adverse Event | 0 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 11 | 12
Not completed — Protocol Violation | 0 | 2
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Peg-IFN + RBV | Arm 2: BOC + Peg-IFN + RBV | Total
Number analyzed (Participants) | 368 | 369 | 737
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (12.0) | 42.4 (12.4) | 43.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 148 | 315
  Male | 201 | 221 | 422

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) 24 Weeks After Completing Study Treatment (SVR24)
Description: SVR24 rates were determined for all participants in Arm 1 and Arm 2. HCV RNA viral load was determined using the Roche COBAS® AmpliPrep/COBAS® TaqMan HCV Test v1.0, which has a lower limit of quantification of 43 IU/mL.
Time Frame: Up to Week 74
Population: The Full Analysis Set (FAS) consisted of all participants who completed the 4-week peg-IFN + RBV lead-in and who were randomized at Week 4.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: Peg-IFN + RBV | Arm 2: BOC + Peg-IFN + RBV
Number analyzed (Participants) | 368 | 369
Percentage of participants | 86.7 | 88.3
Statistical Analysis 1: Comparison: Arm 1: Peg-IFN + RBV vs Arm 2: BOC + Peg-IFN + RBV; Difference in percentage of participants achieving SVR24; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower bound of the 95% CI of the difference in SVR24 % exceeded -10%; Difference in SVR24% in Arm 2 vs. Arm 1 = 1.7, 95% CI 2-sided [-3.2 to 6.5]

2. Secondary Outcome: Percentage of Participants Who Had Undetectable HCV RNA at Week 4 Achieving SVR24
Description: SVR24 rates were determined for only participants that had undetectable HCV RNA at Week 4 of treatment (Arm 1a and Arm 2a). HCV RNA viral load was determined using the Roche COBAS® AmpliPrep/COBAS® TaqMan HCV Test v1.0, which has a lower limit of quantification of 43 IU/mL.
Time Frame: Up to Week 48
Population: The Full Analysis Set (FAS) consisted of all participants who completed the 4-week peg-IFN + RBV lead-in, who were randomized at Week 4, and also had undetectable HCV RNA at Week 4.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1a: Peg-IFN + RBV 24 Weeks: Participants received an initial 4 week lead-in of peg-IFN + RBV. The subset of participants with undetectable HCV RNA at Week 4 received an additional 20 weeks of peg-IFN + RBV for a total of 24 weeks of peg-IFN + RBV therapy.
- Arm 2a: BOC + Peg-IFN + RBV 24 Weeks: Participants received an initial 4 week lead-in of peg-IFN + RBV. The subset of participants with undetectable HCV RNA at Week 4 received an additional 20 weeks of BOC + peg-IFN + RBV for a total of 24 weeks of BOC (added at Week 4) + peg-IFN + RBV therapy.
Arm/Group | Arm 1a: Peg-IFN + RBV 24 Weeks | Arm 2a: BOC + Peg-IFN + RBV 24 Weeks
Number analyzed (Participants) | 108 | 107
Percentage of participants | 87.0 | 97.2
Statistical Analysis 1: Comparison: Arm 1a: Peg-IFN + RBV 24 Weeks vs Arm 2a: BOC + Peg-IFN + RBV 24 Weeks; Test type: Non-Inferiority or Equivalence — The observed lower bound of the 95% CI for the difference was 2.5% (which exceeds 0) for BOC added to peg-IFN + RBV in contrast to peg-IFN + RBV alone; Difference in SVR24% = 10.3, 95% CI 2-sided [2.5 to 18.1]

ADVERSE EVENTS:
Time Frame: Up to 78 weeks
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The All Participants as Treated (APaT) population includes all participants who received at least one dose of study drug.
Arm/Group | Arm 1: Peg-IFN + RBV | Arm 2: BOC + Peg-IFN + RBV
Serious Adverse Events (participants affected / at risk) | 27/368 | 37/369
Other Adverse Events (participants affected / at risk) | 348/368 | 351/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Peg-IFN + RBV (N=368) | Arm 2: BOC + Peg-IFN + RBV (N=369)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Conjunctival melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Miscarriage of partner (Social circumstances) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Peg-IFN + RBV (N=368) | Arm 2: BOC + Peg-IFN + RBV (N=369)
Anaemia (Blood and lymphatic system disorders) | 169 (219) | 168 (210)
Leukopenia (Blood and lymphatic system disorders) | 39 (66) | 33 (46)
Neutropenia (Blood and lymphatic system disorders) | 109 (194) | 108 (161)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (24) | 24 (28)
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 22 (26)
Abdominal pain upper (Gastrointestinal disorders) | 22 (26) | 14 (18)
Diarrhoea (Gastrointestinal disorders) | 62 (77) | 49 (55)
Dry mouth (Gastrointestinal disorders) | 25 (26) | 26 (28)
Dyspepsia (Gastrointestinal disorders) | 23 (25) | 35 (39)
Nausea (Gastrointestinal disorders) | 100 (117) | 94 (112)
Vomiting (Gastrointestinal disorders) | 46 (68) | 53 (78)
Asthenia (General disorders) | 82 (108) | 74 (90)
Chills (General disorders) | 36 (39) | 26 (32)
Fatigue (General disorders) | 118 (135) | 117 (154)
Influenza like illness (General disorders) | 34 (39) | 35 (48)
Pyrexia (General disorders) | 101 (148) | 148 (243)
Haemoglobin decreased (Investigations) | 24 (29) | 31 (33)
Neutrophil count decreased (Investigations) | 24 (30) | 29 (41)
Decreased appetite (Metabolism and nutrition disorders) | 54 (60) | 53 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (49) | 45 (52)
Myalgia (Musculoskeletal and connective tissue disorders) | 61 (79) | 58 (74)
Dizziness (Nervous system disorders) | 46 (51) | 42 (48)
Dysgeusia (Nervous system disorders) | 65 (69) | 94 (95)
Headache (Nervous system disorders) | 118 (152) | 100 (148)
Anxiety (Psychiatric disorders) | 26 (29) | 14 (14)
Depression (Psychiatric disorders) | 29 (38) | 20 (22)
Insomnia (Psychiatric disorders) | 70 (73) | 53 (57)
Irritability (Psychiatric disorders) | 38 (43) | 28 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (83) | 52 (56)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (36) | 34 (38)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 20 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 72 (76) | 70 (74)
Dry skin (Skin and subcutaneous tissue disorders) | 44 (45) | 41 (41)
Pruritus (Skin and subcutaneous tissue disorders) | 75 (85) | 77 (84)
Rash (Skin and subcutaneous tissue disorders) | 69 (82) | 67 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.